CLINICAL TRIAL: NCT06302335
Title: Intraoperative Irrigation of the Surgical Incision With Povidone-iodine vs Saline Solution in Colorectal Surgeries and Its Effects on the Surgical Site Infection
Brief Title: Povidone-iodine vs Saline Solution in Colorectal Surgeries and Its Effects on the Surgical Site Infection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0442
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Surgical Site Infection
Keywords: surgical site infection; colorectal surgey
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This a randomized clinical trial involving patients undergoing colorectal surgeries who will submitted to the application of povidone-iodine versus saline solution in their surgical sites.
Who Masked: Participant
Masking Description: Participants will not know what kind of substance will be used during the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone-iodine arm (Experimental): Patients submitted to colorectal resections using Povidone-iodine in the surgical wound.
  Interventions: Drug: Povidone-iodine
- Saline solution arm. (Active Comparator): Patients submitted to colorectal resections using saline solution in the surgical wound.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Povidone-iodine — Application of Povidone-iodine to the surgical wound of patients submitted to colorectal resections.
  Arms: Povidone-iodine arm
Drug: Saline solution — Application of saline solution to the surgical wound of patients submitted to colorectal resections.
  Arms: Saline solution arm.

SUMMARY:
Considering the relatively high incidence of surgical site infection (SSI) in colorectal surgery, this trial will compare rates of SSI in patients undergoing colorectal resections followed by surgical wound irrigation with povidone-iodine versus the group of patients undergoing surgical wound irrigation with saline solution. The trial will be conducted in a large university hospital in Southern Brazil.

DETAILED DESCRIPTION:
Patients will be randomized to one of the following intervention groups:

Group 1: intraoperative irrigation/washing of the surgical incision with povidone-iodine (PVP-I); Detail: after aponeurotic synthesis and immediately before cutaneous synthesis, the skin and subcutaneous tissue of the surgical incision will be irrigated and washed abundantly with approximately 500ml (depending on the size of the incision) of povidone-iodine solution (PVP-I). The exact volume to be used will be the minimum volume necessary for abundant and efficient washing of the incision tissues. " Group 2: intraoperative irrigation/washing of the surgical incision with saline solution (NaCl 0.9%); Detail: after aponeurotic synthesis and immediately before cutaneous synthesis, the skin and subcutaneous tissue of the surgical incision will be irrigated and washed abundantly with approximately 500ml (depending on the size of the incision) of saline solution (NaCl 0.9%). The exact volume to be used will be the minimum volume necessary for abundant and efficient washing of the incision tissues.

NOTE: other care routines for participating patients will not be changed by this study. Patients will receive mechanical colon preparation and antibiotic prophylaxis according to routines already in place by the assistant team.

Randomization: the block randomization method will be used (blocks of 4 patients each).

Groups 1 and 2 will be compared with each other regarding the outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 18 years of age diagnosed with benign or malignant colorectal diseases undergoing elective open or video-assisted colectomy or proctectomy (resection) at the Hospital de Clinicas de Porto Alegre - Division of Coloproctology.

Exclusion Criteria:

* age under 18;
* surgery classified as dirty;
* urgent/emergency surgery;
* patients undergoing multi-visceral resections (pelvic exenteration or partial resection of any adjacent organ);
* known allergy to iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection within 30 days from the surgical procedure

SECONDARY OUTCOMES:
Intracavitary surgical infection | 30 days
  Infections within the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Damin, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil